CLINICAL TRIAL: NCT05244551
Title: A Phase 1, Open-Label Study of ABSK061 to Assess Safety, Tolerability, and Pharmacokinetics in Patients With Advanced Solid Tumors
Brief Title: A Study to Assess Safety, Tolerability, and Pharmacokinetics of ABSK061 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABSK061-101
Record Dates: First submitted 2022-01-12; First posted 2022-02-17 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABSK061 (Experimental): Dose escalation of oral ABSK061 will be guided by the Bayesian optimal interval (BOIN) design based on safety data collected until a maximum tolerated dose (MTD) or maximum administered dose (MAD) has been identified. During the dose escalation part of the study, patients will receive a single dose of ABSK061 on C1D1 only, and then BID dosing for the rest of the days of cycle 1 and in the subsequent cycles. If the actual elimination half-life of ABSK061 is greatly exceeding that predicted, a run-in period with a single-dose and a longer drug-free observation period could be performed in subsequent patients after the Investigator and Sponsor have discussed and agreed.
  Interventions: Drug: ABSK061

INTERVENTIONS:
Drug: ABSK061 — In the escalation part, patients will receive a single dose of oral ABSK061 on C1D1 only, and then BID dosing for the rest of the days of cycle 1 and in subsequent cycles (28-day cycles). The starting dose is 5 mg BID. In the expansion part, patients will each receive oral ABSK061 at the RDE in repeated 28-day cycles.

SUMMARY:
This is an open-label phase 1 study with expansion. The study will start with a dose escalation of single-agent ABSK061 administered in repeated 28-day cycles in patients with advanced solid tumors to evaluate safety and tolerability. The expansion part will investigate oral ABSK061 at the recommended dose for expansion (RDE) to further evaluate safety and tolerability among selected tumor types. Preliminary antitumor activity will also be assessed.

DETAILED DESCRIPTION:
Escalation Part:

Dose escalation of oral ABSK061 will be guided by the Bayesian optimal interval (BOIN) design based on safety data collected until a maximum tolerated dose (MTD) or maximum administered dose (MAD) has been identified. During the dose escalation part of the study, patients will receive a single dose of ABSK061 on C1D1 only, and then BID dosing for the rest of the days of cycle 1 and in the subsequent cycles. If the actual elimination half-life of ABSK061 is greatly exceeding that predicted, a run-in period with a single-dose and a longer drug-free observation period could be performed in subsequent patients after the Investigator and Sponsor have discussed and agreed.

Expansion Part:

When health authorities outside US require safety data in local population be provided prior to expansion part, a minimum of 3 local subjects will be enrolled and treated at the selected RDE dose level first in that country/region to evaluate the tolerability of ABSK061. The inclusion and exclusion criteria for escalation part will apply for these subjects. After similar safety and tolerability of ABSK061 in patients in the relevant locality have been confirmed by local Investigators and the Sponsor, additional patients will be allowed to enroll in the expansion part.

ELIGIBILITY:
Inclusion Criteria:

1. Patient should understand, sign, and date the written informed consent form prior to screening.
2. Male or female age 18 years or older.
3. For escalation part: patients with histologically confirmed solid tumors who have progressed on or are intolerant of standard therapy or for whom no standard therapy exists.

For expansion Part:

1. Patients with histologically confirmed urothelial carcinoma or cholangiocarcinoma who have progressed on or are intolerant of standard therapy or for whom no standard therapy exists.
2. Patients must have tumors with following FGFR2/3 genetic alterations based on central laboratory test or existing test reports: Urothelial carcinoma: FGFR2/3 fusions and FGFR3 activating mutations Cholangiocarcinoma: FGFR2 fusions and/or arrangements
3. Patients must have at least one measurable target lesion according to RECIST 1.1.
4. Patients are willing to undergo biopsy if archival tumor tissue is not available or the archival specimen deemed inadequate or confirmed FGFR2/3 alterations from existing reports is not available.

4. ECOG performance status 0 or 1 5. Life expectancy ≥3 months 6. Adequate organ function and bone marrow function as indicated by the following screening assessments performed within 14 days prior to the first dose of study drug:

1. Absolute neutrophil count (ANC) ≥1.5×109/L
2. Platelet count (PLT) ≥ 100×109/L without transfusion requirement within 14 days before 1st dose
3. Hemoglobin (Hb)≥90 g/L
4. Total bilirubin (TBIL) ≤1×ULN
5. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5×ULN.
6. Serum creatinine (Cr) of ≤1.5×ULN for the reference laboratory or creatinine clearance (Crcl) ≥ 50 mL/min based on Cockcroft-Gault formula

Exclusion Criteria:

1. Known allergy or hypersensitivity to any component of the investigational product
2. For expansion part only: Previous treatment with FGFR pathway inhibitors or multi-kinase inhibitors which target FGFR inhibition (recommend to consult with sponsor)
3. Has a known additional malignancy that is progressing or has required active treatment.
4. Inability to take oral medication or significant nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude adequate absorption of oral medication
5. Previous anti-cancer therapy, including chemotherapy (chemotherapy with nitrosourea or mitomycin should be at least 6 weeks prior to initiation of study treatment), radiotherapy, molecular targeted therapy or other investigational drugs received ≤4 weeks; endocrine therapy ≤2 weeks or ≤5-half life (whichever is shorter) prior to initiation of study treatment.
6. Major surgery within 4 weeks of the first dose of study drug. Note that all surgical wounds must be healed and free of infection or dehiscence.
7. Prior toxicities from chemotherapy, radiotherapy, and other anti-cancer therapies, including immunotherapy that have not regressed to Grade ≤1 severity (CTCAE V5.0) with the exception of alopecia and vitiligo.
8. Concomitant use of the drugs/remedies that may cause pharmacokinetic drug-drug interactions; consumption of grapefruit juice, grapefruit hybrids, pomegranates, starfruit, pomelos, Seville oranges or juice products within 7 days prior to the first dose of study medication.
9. Active central nervous system (CNS) metastases including presence of cerebral edema, requirement for systemic steroid treatment, disease progression due to intracranial lesions, leptomeningeal metastasis, and other clinical symptoms related to CNS metastases.
10. Impaired cardiac function or clinically significant cardiac disease, including any one of the following:

    * New York Heart Association class III or IV heart disease, active ischemia or any other uncontrolled cardiac condition such as angina pectoris, clinically significant cardiac arrhythmia requiring therapy, uncontrolled hypertension or congestive heart failure
    * Baseline prolongation of the rate-corrected QT interval based on repeated demonstration of QTcF >470 ms or history of long QT interval corrected (QTc) syndrome (Note: QTc interval corrected by Fridericia's formula).
    * Left ventricular ejection fraction (LVEF) <50% or below the institutional lower limit of normal (whichever is higher)
11. Known human immunodeficiency virus (HIV) or active hepatitis B, or active hepatitis C infection; positive tests for hepatitis B virus surface antigen (HBsAg), or antibody to hepatitis B core Ag (HBcAb), or hepatitis C RNA in serum (subjects with history of hepatitis C infection but negative hepatitis C virus polymerase chain reaction (PCR) test are allowed; positive tests for HBV HBsAg or HBcAb with HBV-DNA measurements lower than 1000IU/ml can be included)
12. Any of the following ophthalmological criteria:

    * Current evidence or previous history of retinal pigmented epithelial detachment (RPED)
    * Previous laser treatment or intra-ocular injection for treatment of macular degeneration
    * Current evidence or previous history of dry or wet age-related macular degeneration
    * Current evidence or previous history of retinal vein occlusion (RVO)
    * Current evidence or previous history of retinal degenerative diseases (eg, hereditary)
    * Current evidence or previous history of any other clinically relevant chorioretinal defect
    * Current evidence or previous history of corneal pathology such as conjunctivitis, keratopathy, corneal abrasion or ulceration
13. Patients with refractory/uncontrolled ascites or pleural effusion.
14. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test within 7 days prior to the start of study drug.
15. Non-surgically sterilized male or female patients of childbearing potential must agree to use highly effective methods of birth control during the study and for up to 6 months after the last dose of study drug.
16. Sexually active males, unless they use a condom during intercourse while taking drug and for 5 consecutive compound half-lives plus 60 days after stopping study drug, should not father a child. A condom is required to be used also by vasectomized men to prevent delivery of the drug via seminal fluid.
17. Vaccination with a live, attenuated vaccine within 4 weeks of the first dose of study treatment and while on trial is prohibited except for administration of inactivate vaccines (e.g., COVID-19 vaccines, inactivated influenza vaccines).
18. Any other clinically significant comorbidities, such as uncontrolled pulmonary disease, active infection, or any other condition, which in the judgment of the Investigator, could compromise compliance with the protocol, interfere with the interpretation of study results, or predispose the patient to safety risks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLT | At the end of Cycle 1 (each cycle is 28 days)
  dose-limiting toxicities (DLTs)
Incidence and severity of adverse events (AEs) | Through study completion, an average of half year
  adverse events (AEs), adverse events of special interest (AESIs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Cmax | Through the study completion, an average of half year
  maximum observed concentration
Tmax | Through the study completion, an average of half year
  time to maximum observed concentration
AUC | Through the study completion, an average of half year
  area under the concentration-time curve
t1/2 | Through the study completion, an average of half year
  half-life
Vz/F | Through the study completion, an average of half year
  apparent volume of distribution
CL/F | Through the study completion, an average of half year
  apparent oral clearance
Css_max | Through the study completion, an average of half year
  maximum observed concentration of steady-state
Css_min | Through the study completion, an average of half year
  minimum observed concentration of steady/state
AUCss | Through the study completion, an average of half year
  area under the concentration-time curve of steady/state
Rac | Through the study completion, an average of half year
  accumulation rate
ORR | Through the study completion, an average of half year
  Overall response rate
DoR | Through the study completion, an average of half year
  Duration of response
DCR | from onset of PR or CR to disease progression (up to 100 months)
  Disease control rate
DoR | at 24 weeks
  Duration of response
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Progression-free survival

CONTACTS AND LOCATIONS:
Locations (22):
- Mary Crowley Cancer Research, Dallas, Texas, United States
- China (21):
  - Yuan LU, Shanghai, Abbisko Therapeutics Co., Ltd. 12B Floor, Building 1, Lane 515
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chongqing Daping Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Zhejiang Cancer Hospital, Hangzhou, Gongshu District
  - Sun Yat-sen Memorial Hospital/ the Second Affiliated Hospital of Sun Yat-sen University, Guanzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Xuzhou Center Hospital, Xuzhou, Jiangsu
  - First Hospital of Jilin University, Changchun, Jilin
  - JILIN Cancer Hospital, Changchun, Jilin
  - Yunnan Cancer Hospital, Yunnan, Kunming
  - Liaoning Province Cancer Hospital, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Chongqing University Cancer Hospital, Chongqing, Sichuan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hanzhou, Zhejiang